CLINICAL TRIAL: NCT00421954
Title: Open-label Feasibility Study for the Treatment of Psychotic Adolescents With Ziprasidone in the Inpatient and Day Hospital Settings
Brief Title: Open-label Ziprasidone Study for Psychosis Treatment in Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: # 5239
Record Dates: First submitted 2007-01-12; First posted 2007-01-15 (Estimated); Results first posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Schizophreniform Disorder; Schizoaffective Disorder; Psychosis; Depressive Disorder, Major; Bipolar Disorder
Keywords: psychosis NOS; MDD w/ psychotic features; bipolar disorder w. psychotic features
MeSH Terms: conditions — Psychotic Disorders; Depressive Disorder, Major; Bipolar Disorder; Mental Disorders | interventions — ziprasidone

ARMS (1):
- Ziprasidone (Experimental)
  Interventions: Drug: Ziprasidone

INTERVENTIONS:
Drug: Ziprasidone — subjects will use ziprasidone

SUMMARY:
This open-label study will assess the medication Geodon® (Ziprasidone) in pediatric patients, aged 13-17, diagnosed with psychotic disorder. Eligible adolescents will receive Geodon® for 7 weeks and stay at the NYSPI Children's Day Unit (CDU) during the day. If clinically appropriate, they may also stay at the New York State Psychiatric Institute (NYSPI) Schizophrenia Research Unit (SRU) inpatient facility.

DETAILED DESCRIPTION:
This study is an open-label assessment of the feasibility of treating adolescents with psychotic disorders (schizophreniform disorder, schizoaffective disorder, psychosis not otherwise specified [NOS], major depressive disorder with psychotic features, and bipolar disorder with psychotic features) in an inpatient and day hospital setting with ziprasidone (Geodon). Ziprasidone is a second-generation antipsychotic (SGA) that is FDA-approved for the treatment of schizophrenia and for the treatment of the manic phase of bipolar disorder in adults. It is also used clinically in the treatment of psychotic disorders in children, adolescents and adults. This protocol will help to elucidate the feasibility of studying the treatment of psychotic disorders with ziprasidone in adolescents 13-17 years and help facilitate the further study of the treatment of psychosis with novel agents that have a favorable side effect and weight gain profile.

The duration of the study can be up to 7 weeks. Depending on the level of symptom severity patients will be managed on either the Schizophrenia Research Unit (SRU) (GAS<35, CGI-S>5), or the Children's Day Unit (CDU) of the NYSPI. The seven weeks would encompass a 3 day period at the beginning of the study including time for screening and reviewing lab results. Over a period of one to two weeks patients will be titrated up to 120 mg/day (80 mg for patients under 45kg), and, if necessary, cross tapered off of another SGA that had not been working successfully. Subjects who do not respond to the medication after 1 week at the target dose will be discontinued from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Children who meet DSM-IV criteria for the following psychotic disorders: schizophreniform disorder, schizoaffective disorder, psychosis NOS, major depressive disorder with psychotic features, and bipolar disorder with psychotic features.
2. Children with an IQ of at least 70.
3. Children who are in good physical health.
4. The parent/guardian of the child must be willing to attend all study visits.

Exclusion Criteria:

1. Children who are currently receiving an effective treatment without detrimental side effects.
2. Children who are allergic to Geodon®.
3. Children who have previously failed to respond to an adequate trial of Geodon®.
4. Females who are pregnant or breast-feeding.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2006-05; Primary Completion 2008-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A Maayan, MD, Principal Investigator — NYSPI
Locations (1):
- NYSPI, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: P.I. has left the institution and NYSPI has no access to the data. Results will not be analyzed or presented.
Period: Overall Study
Arm/Group | Ziprasidone
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: P.I. has left the institution and NYSPI has no access to the data. Results will not be analyzed or presented.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Gender
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Weight Gain and Other Side Effects
Time Frame: couple of months
Population: P.I. has left the institution and NYSPI has no access to the data. Results will not be analyzed or presented.
Arm/Group | Ziprasidone
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: P.I. has left the institution and NYSPI has no access to the data. Results will not be analyzed or presented.
Arm/Group | Ziprasidone
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes